CLINICAL TRIAL: NCT02331875
Title: Open Label Single Arm Phase Ib-II Study of Pre-operative IPH2201 in Patients With Locally Advanced Resectable Squamous Cell Carcinoma of the Oral Cavity
Brief Title: Efficacy Study of Pre-operative IPH2201 in Patients With Squamous Cell Carcinoma of the Oral Cavity
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPH2201-201; 2014-002135-34 (EudraCT Number)
Record Dates: First submitted 2015-01-02; First posted 2015-01-06 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

ARMS (1):
- single arm (Experimental): IPH2201 followed by standard surgery and standard postsurgical adjuvant therapy
  Interventions: Drug: IPH2201; Procedure: Standard Surgery; Radiation: Postsurgical Adjuvant Therapy

INTERVENTIONS:
Drug: IPH2201 — The first 6 patients will receive IPH2201, IV, at a dose of 4 mg/kg q2w x 4. Subsequent patients will be treated at a dose of 10 mg/kg q2w x 4.
Procedure: Standard Surgery — After the end of treatment with IPH2201, according to standard recommendations in the relevant country .
Radiation: Postsurgical Adjuvant Therapy — After the standard surgery, according to standard recommendations in the relevant country

SUMMARY:
The primary objective of this open label Phase Ib/II trial is to evaluate the clinical and pharmacological activity of IPH2201 as a single-agent in treatment-naïve pre-operative patients with operable Squamous Cell Carcinoma of the Oral Cavity .

43 patients are planned to be enrolled. The first 6 patients will receive IPH2201 at a dose of 4 mg/kg q2w x 4. Subsequent patients will be treated at a dose of 10 mg/kg q2w x 4. Standard loco-regional treatment with surgery followed by adjuvant therapy will be initiated after the last administration of IPH2201.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed, primary, previously untreated, resectable squamous cell carcinoma of the oral cavity considered clinically and radiologically as intermediate or high risk, classified II ( with large (≥ 3 cm and ≤ 4cm) cT2cN0cM0 tumors or any cT2cN0cM0 tumor invading neighboring structures) III or IVa according to the American Joint Committee on Cancer
* Adequate liver and renal function

Exclusion criteria:

* Other malignancy
* Abnormal cardiac status
* Autoimmune disease
* Serious concurrent uncontrolled medical disorder
* Systemic treatment with corticosteroids or other immunosuppressive agents within 30 days prior to IPH2201 first administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
best objective response rate | 8 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Charité University Medicine Berlin, Berlin, Germany
- Spain (2):
  - Instituto Catalan de Oncologia - L'Hospitalet, L'Hospitalet de Llobregat Barcelona, Spain
  - Hospital Universitario La Paz, Madrid